CLINICAL TRIAL: NCT01920711
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of LCZ696 Compared to Valsartan, on Morbidity and Mortality in Heart Failure Patients (NYHA Class II-IV) With Preserved Ejection Fraction (PARAGON-HF)
Brief Title: Efficacy and Safety of LCZ696 Compared to Valsartan, on Morbidity and Mortality in Heart Failure Patients With Preserved Ejection Fraction
Acronym: PARAGON-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696D2301; 2013-001747-31 (EudraCT Number)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure; preserved ejection fraction; diastolic heart failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCZ696 (Experimental): Single Blind Run-in Period (3-8 weeks): Patients will start on Valsartan 80 mg b.i.d. for 1-2 weeks followed by LCZ696 100 mg b.i.d. for 2-4 weeks prior to randomization into the Double Blind period (up to 57 months). Patients can only be randomized from the run-in period if they meet all of the run-in safety criteria. Target dose of LCZ696 during the double blind period is 200 mg b.i.d.
  Interventions: Drug: LCZ696
- Valsartan (Active Comparator): Single Blind Run-in Period (3-8 weeks): Patients will start on Valsartan 80 mg b.i.d. for 1-2 weeks followed by LCZ696 100 mg b.i.d. for 2-4 weeks prior to randomization into the Double Blind period (up to 57 months). Patients can only be randomized from the run-in period if they meet all of the run-in safety criteria. Target dose of Valsartan during the double blind period is 160 mg b.i.d.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: LCZ696 — LCZ696 50mg, 100mg and 200 mg dosage strengths will be available for dose adjustments.
  Arms: LCZ696
Drug: Valsartan — Valsartan 40mg, 80mg and 160mg dosage strengths will be available for dose adjustments.
  Arms: Valsartan

SUMMARY:
The purpose of this study was to evaluate the effect of LCZ696 compared to valsartan in the reduction of cardiovascular death and heart failure(HF) hospitalizations in patients with HF with preserved ejection fraction.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, parallel group, active-controlled, study to evaluate the efficacy and safety of sacubitril/valsartan compared to valsartan, on morbidity and mortality in heart failure patients (NYHA Class II-IV) with preserved ejection fraction. Specifically, the study evaluated the effect of sacubitril/valsartan compared to the active comparator valsartan in the reduction of the rate of CV death and total HF hospitalizations in patients with HFpEF. The trial consisted of two periods: (1) a single-blind treatment run-in epoch that lasted from 3 to 8 weeks, in which patients received valsartan 80 mg bid, followed by sacubitril/valsartan 100 mg bid and (2) a double-blind randomized treatment epoch (sacubitril/valsartan 200 mg bid or valsartan 160 mg bid). In this study, investigators were responsible for assessing and submitting all events which could potentially fulfill the criteria for the primary, secondary, or other clinical endpoints to a Clinical Endpoint Committee (CEC). Investigator reported events were assessed by the CEC for adjudication.

For angioedema or angioedema-like events, investigators completed an Adjudication Questionnaire for an Angioedema-like Event form. All angioedema reports were forwarded to an Angioedema Adjudication Committee (AAC) by Novartis for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction (LVEF) ≥45% by echo during screening epoch or within 6 months prior to study entry.
* Symptom(s) of heart failure (HF) and requiring treatment with diuretic(s) for HF at least 30 days prior to study entry.
* Current symptom(s) of HF (NYHA class II-IV)
* Structural heart disease (left atrial enlargement or left ventricular hypertrophy) documented by echocardiogram.
* Elevated NT-proBNP

Exclusion Criteria:

* Any prior measurement of LVEF < 40%.
* Acute coronary syndrome (including MI), cardiac surgery, other major CV surgery within 3 months , or urgent percutaneous coronary intervention within 3 months or and elective PCI within 30 days prior to entry.
* Any clinical event within the 6 months prior to entry could have reduced the LVEF (e.g., MI, CABG), unless an echo measurement performed after the event confirms a LVEF ≥45%.
* Current acute decompensated HF requiring therapy.
* Patients who require treatment with 2 or more of the following: an angiotensin converting enzyme inhibitor (ACEI), an angiotensin receptor blocker (ARB) or a renin inhibitor.
* Alternative reason for shortness of breath such as: significant pulmonary disease or severe COPD, hemoglobin (Hgb) <10 g/dl, or body mass index (BMI) > 40 kg/m2.
* Systolic blood pressure (SBP) ≥ 180 mmHg at entry, or SBP >150 mmHg and <180 mmHg at entry unless the patient is receiving 3 or more antihypertensive drugs, or SBP < 110 mmHg at entry.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4822 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (581):
- United States (95):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, West Haven, Connecticut
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Lake Worth, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Covington, Georgia
  - Novartis Investigative Site, Cumming, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Evanston, Illinois
  - Novartis Investigative Site, Hazel Crest, Illinois
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, Maywood, Illinois
  - Novartis Investigative Site, Oakbrook Terrace, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Quincy, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Biddeford, Maine
  - Novartis Investigative Site, Portland, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Grand Blanc, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Cloud, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Kalispell, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Flushing, New York
  - Novartis Investigative Site, Kingston, New York
  - Novartis Investigative Site, Northport, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Saratoga Springs, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Yardley, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Warwick, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, White River Junction, Vermont
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (16):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Australia (5):
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Bundoora, Victoria
  - Novartis Investigative Site, Epping, Victoria
  - Novartis Investigative Site, Geelong, Victoria
- Austria (6):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Grossgmain
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (12):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, De Pinte
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Ottignies
- Brazil (12):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Campina Grande do Sul, Paraná
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Liberdade, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (11):
  - Novartis Investigative Site, Smolyan, Bulgaria
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Silistra
  - Novartis Investigative Site, Sliven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (14):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Thetford-Mines, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- China (25):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Jilin, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Florida Blanca
- Croatia (4):
  - Novartis Investigative Site, Varaždin, HRV
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zadar
  - Novartis Investigative Site, Zagreb
- Czechia (21):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Ivančice, Czech Republic
  - Novartis Investigative Site, Kladno, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Rožnov pod Radhoštěm, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Policska, CZE
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, Ústí nad Labem, CZE
  - Novartis Investigative Site, CZE
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (7):
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Randers
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Viborg
- Finland (3):
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Tampere
- France (14):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (52):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Eilenburg
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Heidenau
  - Novartis Investigative Site, Heppenheim an der Bergstrasse
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Ingelheim
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Meißen
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Muehldorf Am Inn
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Northeim
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rodgau
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Weyhe
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wittenberg
  - Novartis Investigative Site, Würzburg
- Greece (6):
  - Novartis Investigative Site, Athens, Attica
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (9):
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
- India (15):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Chandīgarh, Haryana
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, New Delhi
- Israel (8):
  - Novartis Investigative Site, Lower Galilee, Israel
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Giborim, Holon
- Italy (25):
  - Novartis Investigative Site, Aosta, AO
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Vimercate, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Ariccia, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Palmanova, UD
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Saronno, Va
  - Novartis Investigative Site, Venezia, VE
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
- Japan (18):
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kan’onjichō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Mexico (10):
  - Novartis Investigative Site, Torreón, Coahulia
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, San Juan del Río, Querétaro
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Querétaro
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (15):
  - Novartis Investigative Site, Apeldoorn, DZ
  - Novartis Investigative Site, The Hague, NL
  - Novartis Investigative Site, Almelo, PP
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Blaricum
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
- Norway (4):
  - Novartis Investigative Site, Loerenskog
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Tromsø
- Peru (5):
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
- Philippines (3):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Quezon City
- Poland (13):
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Sandomierz
  - Novartis Investigative Site, Staszów
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Warszawa/Anin
  - Novartis Investigative Site, Zabrze
  - Novartis Investigative Site, Zamość
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Romania (10):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Sibiu, Jud. Iasi
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (14):
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Serbia (3):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Niška Banja
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (18):
  - Novartis Investigative Site, Brezno, Slovak Republic
  - Novartis Investigative Site, Komárno, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Námestovo, Slovak Republic
  - Novartis Investigative Site, Považská Bystrica, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Trebišov
  - Novartis Investigative Site, Žilina
- Slovenia (2):
  - Novartis Investigative Site, Golnik
  - Novartis Investigative Site, Ljubljana
- South Africa (10):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Alberton
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Tongaat
  - Novartis Investigative Site, Western Cape
  - Novartis Investigative Site, Worcester
- South Korea (9):
  - Novartis Investigative Site, Gyeonggi-do, Bucheon Si
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Incheon, KOR
  - Novartis Investigative Site, Seoul, KOR
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Spain (24):
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Aranda de Duero, Castille and León
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Olot, Girona
  - Novartis Investigative Site, Móstoles, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Ciudad Real
  - Novartis Investigative Site, Madrid
- Sweden (8):
  - Novartis Investigative Site, Danderyd
  - Novartis Investigative Site, Falun
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Karlstad
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Västerås
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Biel
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Taiwan (8):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Yilan
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Haydarpasa Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Sivas
- United Kingdom (29):
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Stockton-on-Tees, Cleveland
  - Novartis Investigative Site, Darlington, Co Durham
  - Novartis Investigative Site, Durham, County Durham
  - Novartis Investigative Site, Torquay, Devon
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Peterborough, GBR
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Portsmouth, Hampshire
  - Novartis Investigative Site, Oldham, Lancashire
  - Novartis Investigative Site, Harrow, Middlesex
  - Novartis Investigative Site, Portadown, Nothern Ireland
  - Novartis Investigative Site, Wansford, Peterborough
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Gateshead, Tyne and Wear
  - Novartis Investigative Site, Clydebank, West Dumbartonshire
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Swindon
  - Novartis Investigative Site, Wiltshire
  - Novartis Investigative Site, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Yang M, Henderson AD, Anand IS, Desai AS, Lam CSP, Maggioni AP, Martinez FA, Rouleau JL, Swedberg K, Vaduganathan M, van Veldhuisen DJ, Zannad F, Zile MR, Packer M, Rizkala A, Lewis EF, Jhund PS, Solomon SD, McMurray JJV. Sacubitril/valsartan and quality of life assessed using the EuroQol Five-dimension Three-level questionnaire level sum score (EQ-5D-3L-LSS) in patients with HFrEF and HFmrEF/HFpEF. Eur Heart J Cardiovasc Pharmacother. 2025 Nov 4;11(7):574-589. doi: 10.1093/ehjcvp/pvaf064. PMID 40839760
- [Derived] Lu H, Claggett BL, Minamisawa M, Ostrominski JW, Foa A, Pabon MA, Kalayci A, Vaduganathan M, Cikes M, Shah AM, Desai AS, McMurray JJV, Jhund PS, Packer M, Lefkowitz M, Rouleau JL, Zile MR, Zannad F, Hegde SM, Solomon SD, Skali H. Prognostic Significance of Nutritional Scores in Patients With Heart Failure: Insights From the PARAGON-HF Trial. J Am Heart Assoc. 2025 May 6;14(9):e038872. doi: 10.1161/JAHA.124.038872. Epub 2025 Apr 23. PMID 40265602
- [Derived] Kondo T, Jhund PS, Anand IS, Claggett BL, Desai AS, Docherty KF, Lam CSP, Lefkowitz MP, Maggioni AP, Martinez FA, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, Packer M, Solomon SD, McMurray JJV. Effects of Sacubitril/Valsartan According to Natriuretic Peptide Levels in Patients Enrolled in PARADIGM-HF and PARAGON-HF. JACC Heart Fail. 2025 Jun;13(6):927-939. doi: 10.1016/j.jchf.2024.12.010. Epub 2025 Mar 12. PMID 40088233
- [Derived] Peikert A, Vaduganathan M, Claggett BL, Kulac IJ, Litwin S, Zile M, Desai AS, Jhund PS, Butt JH, Lam CSP, Martinez F, Van Veldhuisen DJ, Zannad F, Rouleau J, Lefkowitz M, McMurray JJV, Solomon SD, Packer M. Near-universal prevalence of central adiposity in heart failure with preserved ejection fraction: the PARAGON-HF trial. Eur Heart J. 2025 Jul 1;46(25):2372-2390. doi: 10.1093/eurheartj/ehaf057. PMID 39873282
- [Derived] Mc Causland FR, Vaduganathan M, Claggett B, Gori M, Jhund PS, McGrath MM, Neuen BL, Packer M, Pfeffer MA, Rouleau JL, Senni M, Swedberg K, Zannad F, Zile M, Lefkowitz MP, McMurray JJV, Solomon SD. Angiotensin Receptor Neprilysin Inhibition and Cardiovascular Outcomes Across the Kidney Function Spectrum: The PARAGON-HF Trial. JACC Heart Fail. 2025 Jan;13(1):105-114. doi: 10.1016/j.jchf.2024.08.022. Epub 2024 Nov 20. PMID 39570234
- [Derived] Lu H, Claggett BL, Packer M, Pfeffer MA, Swedberg K, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund PS, McMurray JJV, Solomon SD, Vaduganathan M. Visit-to-visit changes in heart rate in heart failure: A pooled participant-level analysis of the PARADIGM-HF and PARAGON-HF trials. Eur J Heart Fail. 2025 Jan;27(1):60-68. doi: 10.1002/ejhf.3487. Epub 2024 Oct 22. PMID 39439294
- [Derived] Lu H, Claggett BL, Packer M, Pabon MA, Pfeffer MA, Lewis EF, Lam CSP, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund PS, McMurray JJV, Solomon SD, Vaduganathan M. Race in Heart Failure: A Pooled Participant-Level Analysis of the Global PARADIGM-HF and PARAGON-HF Trials. JACC Heart Fail. 2025 Jan;13(1):58-71. doi: 10.1016/j.jchf.2024.08.008. Epub 2024 Aug 31. PMID 39387766
- [Derived] Lu H, Claggett BL, Packer M, Pfeffer MA, Lam CSP, Zile MR, Desai AS, Jhund P, Lefkowitz M, McMurray JJV, Solomon SD, Vaduganathan M. Sacubitril/valsartan reduces incident anaemia and iron therapy utilization in heart failure: The PARAGON-HF trial. Eur J Heart Fail. 2025 Jan;27(1):85-95. doi: 10.1002/ejhf.3414. Epub 2024 Sep 1. PMID 39217577
- [Derived] Lu H, Chatur S, Lee S, Inciardi RM, Abanda M, Mc Causland FR, Kalayci A, Taheri KK, Shah AM, Cikes M, Claggett BL, Prasad N, Lam CSP, O'Meara E, Wang X, McMurray JJV, Pfeffer MA, Hegde SM, Solomon SD, Skali H. Relationship Between Cardiac Structure and Function With Renal Function Trajectory and Outcomes in Patients With Heart Failure: Insights From the PARAGON-HF Trial. Circ Heart Fail. 2024 Oct;17(10):e011942. doi: 10.1161/CIRCHEARTFAILURE.124.011942. Epub 2024 Aug 30. PMID 39212045
- [Derived] Lu H, Claggett BL, Packer M, Lam CSP, Swedberg K, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund P, McMurray JJV, Solomon SD, Vaduganathan M. Effects of Sacubitril/Valsartan on All-Cause Hospitalizations in Heart Failure: Post Hoc Analysis of the PARADIGM-HF and PARAGON-HF Randomized Clinical Trials. JAMA Cardiol. 2024 Nov 1;9(11):1047-1052. doi: 10.1001/jamacardio.2024.2566. PMID 39210725
- [Derived] Yoon M, Kim W, Kook W, Park JJ, Greenberg B. Analysis of the PARAGON-HF Study Results Using Win Ratio. Circ Heart Fail. 2024 Sep;17(9):e011860. doi: 10.1161/CIRCHEARTFAILURE.124.011860. Epub 2024 Aug 28. PMID 39193709
- [Derived] Lassen MCH, Ostrominski JW, Claggett BL, Packer M, Zile M, Desai AS, Shah AM, Cikes M, Merkely B, Gori M, Wang X, Hegde SM, Pfeffer MA, Lefkowitz M, McMurray JJV, Solomon SD, Vaduganathan M. Cardiovascular-kidney-metabolic overlap in heart failure with preserved ejection fraction: Cardiac structure and function, clinical outcomes, and response to sacubitril/valsartan in PARAGON-HF. Eur J Heart Fail. 2024 Aug;26(8):1762-1774. doi: 10.1002/ejhf.3304. Epub 2024 Jun 26. PMID 38932589
- [Derived] Patel-Murray NL, Zhang L, Claggett BL, Xu D, Serrano-Fernandez P, Healey M, Wandel S, Chen CW, Jacob J, Xu H, Turner GM, Chutkow W, Yates DP, O'Donnell CJ, Prescott MF, Lefkowitz M, Gimpelewicz CR, Beste MT, Zhao F, Gou L, Desai AS, Jhund PS, Packer M, Pfeffer MA, Redfield MM, Rouleau JL, Zannad F, Zile MR, McMurray JJV, Mendelson MM, Solomon SD, Cunningham JW. Aptamer Proteomics for Biomarker Discovery in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Proteomic Substudy. J Am Heart Assoc. 2024 Jul 2;13(13):e033544. doi: 10.1161/JAHA.123.033544. Epub 2024 Jun 21. PMID 38904251
- [Derived] Chatur S, Beldhuis IE, Claggett BL, McCausland FR, Neuen BL, Desai AS, Rouleau JL, Zile MR, Packer M, Pfeffer MA, Lefkowitz MP, McMurray JJV, Solomon SD, Vaduganathan M. Sacubitril/Valsartan in Patients With Heart Failure and Deterioration in eGFR to <30 mL/min/1.73 m2. JACC Heart Fail. 2024 Oct;12(10):1692-1703. doi: 10.1016/j.jchf.2024.03.014. Epub 2024 Jun 5. PMID 38842957
- [Derived] Dewan P, Shen L, Pedro Ferreira J, Jhund PS, Anand IS, Chandra A, Chiang LM, Claggett B, Desai AS, Gong J, Lam CSP, Lefkowitz MP, Maggioni AP, Martinez F, Packer M, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Solomon SD, McMurray JJV. Effect of Sacubitril/Valsartan on Cognitive Function in Patients With Heart Failure With Preserved Ejection Fraction: A Prespecified Analysis of PARAGON-HF. Circulation. 2024 Jul 23;150(4):272-282. doi: 10.1161/CIRCULATIONAHA.124.068774. Epub 2024 Jun 6. PMID 38841854
- [Derived] Foa A, Vaduganathan M, Claggett BL, Pabon MA, Lu H, Pfeffer MA, Packer M, Vardeny O, Rouleau JL, Lefkowitz M, Mentz RJ, Jhund PS, Desai AS, McMurray JJV, Solomon SD. Sacubitril/Valsartan-Related Hypotension in Patients With Heart Failure and Preserved or Mildly Reduced Ejection Fraction. J Am Coll Cardiol. 2024 May 7;83(18):1731-1739. doi: 10.1016/j.jacc.2024.02.035. Epub 2024 Mar 25. PMID 38537919
- [Derived] Bhatt AS, Vaduganathan M, Claggett BL, Kulac IJ, Anand IS, Desai AS, Fang JC, Hernandez AF, Jhund PS, Kosiborod MN, Sabatine MS, Shah SJ, Vardeny O, McMurray JJV, Solomon SD, Gaziano TA. Cost Effectiveness of Dapagliflozin for Heart Failure Across the Spectrum of Ejection Fraction: An Economic Evaluation Based on Pooled, Individual Participant Data From the DELIVER and DAPA-HF Trials. J Am Heart Assoc. 2024 Mar 5;13(5):e032279. doi: 10.1161/JAHA.123.032279. Epub 2024 Feb 23. PMID 38390793
- [Derived] Butt JH, Jering K, DE Boer RA, Claggett BL, Desai AS, Hernandez AF, Inzucchi SE, Jhund PS, Kober L, Kosiborod MN, Lam CSP, Martinez FA, Ponikowski P, Sabatine MS, Shah SJ, Vaduganathan M, Langkilde AM, Bengtsson O, Petersson M, Sjostrand M, Wilderang U, Solomon SD, McMurray JJV. Heart Failure, Investigator-Reported Sleep Apnea and Dapagliflozin: A Patient-Level Pooled Meta-Analysis of DAPA-HF and DELIVER. J Card Fail. 2024 Mar;30(3):436-448. doi: 10.1016/j.cardfail.2023.08.027. Epub 2023 Dec 15. PMID 38104937
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Kondo T, Jering KS, Jhund PS, Anand IS, Desai AS, Lam CSP, Maggioni AP, Martinez FA, Packer M, Petrie MC, Pfeffer MA, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Solomon SD, McMurray JJV. Predicting Stroke in Heart Failure and Preserved Ejection Fraction Without Atrial Fibrillation. Circ Heart Fail. 2023 Jul;16(7):e010377. doi: 10.1161/CIRCHEARTFAILURE.122.010377. Epub 2023 Jun 23. PMID 37350280
- [Derived] Inciardi RM, Abanda M, Shah AM, Cikes M, Claggett B, Skali H, Vaduganathan M, Prasad N, Litwin S, Merkely B, Kosztin A, Nagy KV, Shah SJ, Mullens W, Zile MR, Lam CSP, Pfeffer MA, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Right Ventricular Function and Pulmonary Coupling in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2023 Aug 8;82(6):489-499. doi: 10.1016/j.jacc.2023.05.010. Epub 2023 May 22. PMID 37225045
- [Derived] Lyu T, Bornkamp B, Mueller-Velten G, Schmidli H. Bayesian inference for a principal stratum estimand on recurrent events truncated by death. Biometrics. 2023 Dec;79(4):3792-3802. doi: 10.1111/biom.13831. Epub 2023 Jan 30. PMID 36647690
- [Derived] Curtain JP, Adamson C, Kondo T, Butt JH, Desai AS, Zannad F, Rouleau JL, Rohde LE, Kober L, Anand IS, van Veldhuisen DJ, Zile MR, Lefkowitz MP, Solomon SD, Packer M, Petrie MC, Jhund PS, McMurray JJV. Investigator-reported ventricular arrhythmias and mortality in heart failure with mildly reduced or preserved ejection fraction. Eur Heart J. 2023 Feb 21;44(8):668-677. doi: 10.1093/eurheartj/ehac801. PMID 36632831
- [Derived] Butt JH, Dewan P, Jhund PS, Anand IS, Atar D, Ge J, Desai AS, Echeverria LE, Kober L, Lam CSP, Maggioni AP, Martinez F, Packer M, Rouleau JL, Sim D, Van Veldhuisen DJ, Vrtovec B, Zannad F, Zile MR, Gong J, Lefkowitz MP, Rizkala AR, Solomon SD, McMurray JJV. Sacubitril/Valsartan and Frailty in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2022 Sep 20;80(12):1130-1143. doi: 10.1016/j.jacc.2022.06.037. Epub 2022 Aug 29. PMID 36050227
- [Derived] Chatur S, Vaduganathan M, Peikert A, Claggett BL, McCausland FR, Skali H, Pfeffer MA, Beldhuis IE, Kober L, Seferovic P, Lefkowitz M, McMurray JJV, Solomon SD. Longitudinal trajectories in renal function before and after heart failure hospitalization among patients with heart failure with preserved ejection fraction in the PARAGON-HF trial. Eur J Heart Fail. 2022 Oct;24(10):1906-1914. doi: 10.1002/ejhf.2638. Epub 2022 Aug 15. PMID 35895867
- [Derived] Wijkman MO, Claggett B, Vaduganathan M, Cunningham JW, Rorth R, Jackson A, Packer M, Zile M, Rouleau J, Swedberg K, Lefkowitz M, Shah SJ, Pfeffer MA, McMurray JJV, Solomon SD. Effects of sacubitril/valsartan on glycemia in patients with diabetes and heart failure: the PARAGON-HF and PARADIGM-HF trials. Cardiovasc Diabetol. 2022 Jun 18;21(1):110. doi: 10.1186/s12933-022-01545-1. PMID 35717169
- [Derived] Vaduganathan M, Claggett BL, Inciardi RM, Fonarow GC, McMurray JJV, Solomon SD. Estimating the Benefits of Combination Medical Therapy in Heart Failure With Mildly Reduced and Preserved Ejection Fraction. Circulation. 2022 Jun 7;145(23):1741-1743. doi: 10.1161/CIRCULATIONAHA.121.058929. Epub 2022 May 23. No abstract available. PMID 35603667
- [Derived] Vaduganathan M, Claggett BL, McMurray JJV, Solomon SD. Health Status Trajectories Before and After Hospitalization for Heart Failure. Circulation. 2022 Jun 21;145(25):1872-1874. doi: 10.1161/CIRCULATIONAHA.122.059282. Epub 2022 May 21. No abstract available. PMID 35603665
- [Derived] Cikes M, Planinc I, Claggett B, Cunningham J, Milicic D, Sweitzer N, Senni M, Gori M, Linssen G, Shah SJ, Packer M, Pfeffer M, Zile MR, Anand I, Chiang LM, Lam CSP, Redfield M, Desai AS, McMurray JJV, Solomon SD. Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. JACC Heart Fail. 2022 May;10(5):336-346. doi: 10.1016/j.jchf.2022.01.018. Epub 2022 Apr 6. PMID 35483796
- [Derived] Jackson AM, Rorth R, Liu J, Kristensen SL, Anand IS, Claggett BL, Cleland JGF, Chopra VK, Desai AS, Ge J, Gong J, Lam CSP, Lefkowitz MP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rizkala AR, Rouleau JL, Seferovic PM, Tromp J, Van Veldhuisen DJ, Yilmaz MB, Zannad F, Zile MR, Kober L, Petrie MC, Jhund PS, Solomon SD, McMurray JJV; PARAGON-HF Committees and Investigators. Diabetes and pre-diabetes in patients with heart failure and preserved ejection fraction. Eur J Heart Fail. 2022 Mar;24(3):497-509. doi: 10.1002/ejhf.2403. Epub 2022 Jan 4. PMID 34918855
- [Derived] Desai AS, Vaduganathan M, Cleland JG, Claggett BL, Barkoudah E, Finn P, McCausland FR, Yilmaz MB, Lefkowitz M, Shi V, Pfeffer MA, McMurray JJV, Solomon SD. Mode of Death in Patients With Heart Failure and Preserved Ejection Fraction: Insights From PARAGON-HF Trial. Circ Heart Fail. 2021 Dec;14(12):e008597. doi: 10.1161/CIRCHEARTFAILURE.121.008597. Epub 2021 Nov 22. PMID 34807713
- [Derived] Mooney L, Hawkins NM, Jhund PS, Redfield MM, Vaduganathan M, Desai AS, Rouleau JL, Minamisawa M, Shah AM, Lefkowitz MP, Zile MR, Van Veldhuisen DJ, Pfeffer MA, Anand IS, Maggioni AP, Senni M, Claggett BL, Solomon SD, McMurray JJV. Impact of Chronic Obstructive Pulmonary Disease in Patients With Heart Failure With Preserved Ejection Fraction: Insights From PARAGON-HF. J Am Heart Assoc. 2021 Dec 7;10(23):e021494. doi: 10.1161/JAHA.121.021494. Epub 2021 Nov 19. PMID 34796742
- [Derived] Jackson AM, Jhund PS, Anand IS, Dungen HD, Lam CSP, Lefkowitz MP, Linssen G, Lund LH, Maggioni AP, Pfeffer MA, Rouleau JL, Saraiva JFK, Senni M, Vardeny O, Wijkman MO, Yilmaz MB, Saito Y, Zile MR, Solomon SD, McMurray JJV. Sacubitril-valsartan as a treatment for apparent resistant hypertension in patients with heart failure and preserved ejection fraction. Eur Heart J. 2021 Sep 21;42(36):3741-3752. doi: 10.1093/eurheartj/ehab499. PMID 34392331
- [Derived] Felker GM, Butler J, Januzzi JL Jr, Desai AS, McMurray JJV, Solomon SD. Probabilistic Readjudication of Heart Failure Hospitalization Events in the PARAGON-HF Study. Circulation. 2021 Jun 8;143(23):2316-2318. doi: 10.1161/CIRCULATIONAHA.121.054496. Epub 2021 Jun 7. No abstract available. PMID 34097449
- [Derived] Selvaraj S, Claggett BL, Packer M, Zannad F, Anand IS, Pieske B, Zhao Z, Shi VC, Lefkowitz MP, McMurray JJV, Solomon SD. Effects of Sacubitril/Valsartan on Serum Lipids in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2021 Sep 7;10(17):e022069. doi: 10.1161/JAHA.121.022069. Epub 2021 May 16. PMID 33998278
- [Derived] Shen L, Jhund PS, Anand IS, Bhatt AS, Desai AS, Maggioni AP, Martinez FA, Pfeffer MA, Rizkala AR, Rouleau JL, Swedberg K, Vaduganathan M, Vardeny O, van Veldhuisen DJ, Zannad F, Zile MR, Packer M, Solomon SD, McMurray JJV. Incidence and Outcomes of Pneumonia in Patients With Heart Failure. J Am Coll Cardiol. 2021 Apr 27;77(16):1961-1973. doi: 10.1016/j.jacc.2021.03.001. PMID 33888245
- [Derived] Tromp J, Claggett BL, Liu J, Jackson AM, Jhund PS, Kober L, Widimsky J, Boytsov SA, Chopra VK, Anand IS, Ge J, Chen CH, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, Rizkala AR, Inubushi-Molessa A, Lefkowitz MP, Shi VC, McMurray JJV, Solomon SD, Lam CSP; PARAGON-HF Investigators. Global Differences in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. Circ Heart Fail. 2021 Apr;14(4):e007901. doi: 10.1161/CIRCHEARTFAILURE.120.007901. Epub 2021 Apr 19. PMID 33866828
- [Derived] Vaduganathan M, Cunningham JW, Claggett BL, Causland FM, Barkoudah E, Finn P, Zannad F, Pfeffer MA, Rizkala AR, Sabarwal S, McMurray JJV, Solomon S, Desai AS. Worsening Heart Failure Episodes Outside a Hospital Setting in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. JACC Heart Fail. 2021 May;9(5):374-382. doi: 10.1016/j.jchf.2021.01.014. Epub 2021 Apr 7. PMID 33839075
- [Derived] Gronda E, Vanoli E, Iacoviello M. The PARAGON-HF trial: the sacubitril/valsartan in heart failure with preserved ejection fraction. Eur Heart J Suppl. 2020 Nov 18;22(Suppl L):L77-L81. doi: 10.1093/eurheartj/suaa140. eCollection 2020 Nov. PMID 33727901
- [Derived] Jering K, Claggett B, Redfield MM, Shah SJ, Anand IS, Martinez F, Sabarwal SV, Seferovic PM, Kerr Saraiva JF, Katova T, Lefkowitz MP, Pfeffer MA, McMurray JJV, Solomon SD. Burden of Heart Failure Signs and Symptoms, Prognosis, and Response to Therapy: The PARAGON-HF Trial. JACC Heart Fail. 2021 May;9(5):386-397. doi: 10.1016/j.jchf.2021.01.011. Epub 2021 Mar 10. PMID 33714741
- [Derived] Jering KS, Zannad F, Claggett B, Mc Causland FR, Ferreira JP, Desai A, Barkoudah E, McMurray JJV, Pfeffer MA, Solomon SD. Cardiovascular and Renal Outcomes of Mineralocorticoid Receptor Antagonist Use in PARAGON-HF. JACC Heart Fail. 2021 Jan;9(1):13-24. doi: 10.1016/j.jchf.2020.08.014. Epub 2020 Nov 11. PMID 33189633
- [Derived] Mc Causland FR, Lefkowitz MP, Claggett B, Anavekar NS, Senni M, Gori M, Jhund PS, McGrath MM, Packer M, Shi V, Van Veldhuisen DJ, Zannad F, Comin-Colet J, Pfeffer MA, McMurray JJV, Solomon SD. Angiotensin-Neprilysin Inhibition and Renal Outcomes in Heart Failure With Preserved Ejection Fraction. Circulation. 2020 Sep 29;142(13):1236-1245. doi: 10.1161/CIRCULATIONAHA.120.047643. Epub 2020 Aug 17. PMID 32845715
- [Derived] Cunningham JW, Claggett BL, O'Meara E, Prescott MF, Pfeffer MA, Shah SJ, Redfield MM, Zannad F, Chiang LM, Rizkala AR, Shi VC, Lefkowitz MP, Rouleau J, McMurray JJV, Solomon SD, Zile MR. Effect of Sacubitril/Valsartan on Biomarkers of Extracellular Matrix Regulation in Patients With HFpEF. J Am Coll Cardiol. 2020 Aug 4;76(5):503-514. doi: 10.1016/j.jacc.2020.05.072. PMID 32731928
- [Derived] Cunningham JW, Vaduganathan M, Claggett BL, Zile MR, Anand IS, Packer M, Zannad F, Lam CSP, Janssens S, Jhund PS, Kober L, Rouleau J, Shah SJ, Chopra VK, Shi VC, Lefkowitz MP, Prescott MF, Pfeffer MA, McMurray JJV, Solomon SD. Effects of Sacubitril/Valsartan on N-Terminal Pro-B-Type Natriuretic Peptide in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2020 May;8(5):372-381. doi: 10.1016/j.jchf.2020.03.002. Epub 2020 Mar 30. PMID 32241619
- [Derived] Selvaraj S, Claggett BL, Bohm M, Anker SD, Vaduganathan M, Zannad F, Pieske B, Lam CSP, Anand IS, Shi VC, Lefkowitz MP, McMurray JJV, Solomon SD. Systolic Blood Pressure in Heart Failure With Preserved Ejection Fraction Treated With Sacubitril/Valsartan. J Am Coll Cardiol. 2020 Apr 14;75(14):1644-1656. doi: 10.1016/j.jacc.2020.02.009. Epub 2020 Mar 16. PMID 32192799
- [Derived] Shah AM, Cikes M, Prasad N, Li G, Getchevski S, Claggett B, Rizkala A, Lukashevich I, O'Meara E, Ryan JJ, Shah SJ, Mullens W, Zile MR, Lam CSP, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Echocardiographic Features of Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction. J Am Coll Cardiol. 2019 Dec 10;74(23):2858-2873. doi: 10.1016/j.jacc.2019.09.063. PMID 31806129
- [Derived] Solomon SD, Vaduganathan M, L Claggett B, Packer M, Zile M, Swedberg K, Rouleau J, A Pfeffer M, Desai A, Lund LH, Kober L, Anand I, Sweitzer N, Linssen G, Merkely B, Luis Arango J, Vinereanu D, Chen CH, Senni M, Sibulo A, Boytsov S, Shi V, Rizkala A, Lefkowitz M, McMurray JJV. Sacubitril/Valsartan Across the Spectrum of Ejection Fraction in Heart Failure. Circulation. 2020 Feb 4;141(5):352-361. doi: 10.1161/CIRCULATIONAHA.119.044586. Epub 2019 Nov 17. PMID 31736342
- [Derived] McMurray JJV, Jackson AM, Lam CSP, Redfield MM, Anand IS, Ge J, Lefkowitz MP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Rizkala AR, Sabarwal SV, Shah AM, Shah SJ, Shi VC, van Veldhuisen DJ, Zannad F, Zile MR, Cikes M, Goncalvesova E, Katova T, Kosztin A, Lelonek M, Sweitzer N, Vardeny O, Claggett B, Jhund PS, Solomon SD. Effects of Sacubitril-Valsartan Versus Valsartan in Women Compared With Men With Heart Failure and Preserved Ejection Fraction: Insights From PARAGON-HF. Circulation. 2020 Feb 4;141(5):338-351. doi: 10.1161/CIRCULATIONAHA.119.044491. Epub 2019 Nov 17. PMID 31736337
- [Derived] Vaduganathan M, Claggett BL, Desai AS, Anker SD, Perrone SV, Janssens S, Milicic D, Arango JL, Packer M, Shi VC, Lefkowitz MP, McMurray JJV, Solomon SD. Prior Heart Failure Hospitalization, Clinical Outcomes, and Response to Sacubitril/Valsartan Compared With Valsartan in HFpEF. J Am Coll Cardiol. 2020 Jan 28;75(3):245-254. doi: 10.1016/j.jacc.2019.11.003. Epub 2019 Nov 11. PMID 31726194
- [Derived] Solomon SD, McMurray JJV, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Claggett B, Jhund PS, Boytsov SA, Comin-Colet J, Cleland J, Dungen HD, Goncalvesova E, Katova T, Kerr Saraiva JF, Lelonek M, Merkely B, Senni M, Shah SJ, Zhou J, Rizkala AR, Gong J, Shi VC, Lefkowitz MP; PARAGON-HF Investigators and Committees. Angiotensin-Neprilysin Inhibition in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2019 Oct 24;381(17):1609-1620. doi: 10.1056/NEJMoa1908655. Epub 2019 Sep 1. PMID 31475794
- [Derived] Chandra A, Vaduganathan M, Lewis EF, Claggett BL, Rizkala AR, Wang W, Lefkowitz MP, Shi VC, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Health-Related Quality of Life in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. JACC Heart Fail. 2019 Oct;7(10):862-874. doi: 10.1016/j.jchf.2019.05.015. Epub 2019 Jul 10. PMID 31302043
- [Derived] Solomon SD, Rizkala AR, Lefkowitz MP, Shi VC, Gong J, Anavekar N, Anker SD, Arango JL, Arenas JL, Atar D, Ben-Gal T, Boytsov SA, Chen CH, Chopra VK, Cleland J, Comin-Colet J, Duengen HD, Echeverria Correa LE, Filippatos G, Flammer AJ, Galinier M, Godoy A, Goncalvesova E, Janssens S, Katova T, Kober L, Lelonek M, Linssen G, Lund LH, O'Meara E, Merkely B, Milicic D, Oh BH, Perrone SV, Ranjith N, Saito Y, Saraiva JF, Shah S, Seferovic PM, Senni M, Sibulo AS Jr, Sim D, Sweitzer NK, Taurio J, Vinereanu D, Vrtovec B, Widimsky J Jr, Yilmaz MB, Zhou J, Zweiker R, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, McMurray JJV. Baseline Characteristics of Patients With Heart Failure and Preserved Ejection Fraction in the PARAGON-HF Trial. Circ Heart Fail. 2018 Jul;11(7):e004962. doi: 10.1161/CIRCHEARTFAILURE.118.004962. PMID 29980595
- [Derived] Mutze T, Glimm E, Schmidli H, Friede T. Group sequential designs with robust semiparametric recurrent event models. Stat Methods Med Res. 2019 Aug;28(8):2385-2403. doi: 10.1177/0962280218780538. Epub 2018 Jun 11. PMID 29890892
- [Derived] Solomon SD, Rizkala AR, Gong J, Wang W, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, Desai AS, Shi VC, Lefkowitz MP, McMurray JJV. Angiotensin Receptor Neprilysin Inhibition in Heart Failure With Preserved Ejection Fraction: Rationale and Design of the PARAGON-HF Trial. JACC Heart Fail. 2017 Jul;5(7):471-482. doi: 10.1016/j.jchf.2017.04.013. Epub 2017 Jun 26. PMID 28662936
- [Derived] Rossi A, Gheorghiade M, Triposkiadis F, Solomon SD, Pieske B, Butler J. Left atrium in heart failure with preserved ejection fraction: structure, function, and significance. Circ Heart Fail. 2014 Nov;7(6):1042-9. doi: 10.1161/CIRCHEARTFAILURE.114.001276. No abstract available. PMID 25415957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4822 patients were randomized at 755 sites in 43 countries. 2419 participants were randomized into the LCZ696 treatment group and 2403 were randomized into the valsartan treatment group.
Groups:
- LCZ696: Single Blind Run-in Period (3-8 weeks): Prior optional valsartan run-in 40 mg bid for 1-2 weeks for some patients followed by Valsartan 80 mg bid for 1-2 weeks followed by LCZ696 100 mg bid for 2-4 weeks prior to randomization into the Double Blind period (up to 57 months). Patients could only be randomized from the run-in period if they met all of the run-in safety criteria. Target dose of LCZ696 during the double blind period was 200 mg bid
- Valsartan: Single Blind Run-in Period (3-8 weeks): Prior optional valsartan run-in 40 mg bid for 1-2 weeks for some patients, followed by Valsartan 80 mg bid. for 1-2 weeks followed by LCZ696 100 mg bid for 2-4 weeks prior to randomization into the Double Blind period (up to 57 months). Patients could only be randomized from the run-in period if they met all of the run-in safety criteria. Target dose of Valsartan during the double blind period was 160 mg bid
Period: Overall Study
Arm/Group | LCZ696 | Valsartan
Started | 2419 | 2403
Completed | 2055 | 2030
Not Completed | 364 | 373
Not completed — Death | 347 | 356
Not completed — Lost to Follow-up | 13 | 14
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: Randomized set totaled 4822 patients. Full Analysis Set consisted of 4796 patients: primary efficacy population used in the analyses for all efficacy endpoints, includes all randomized patients minus 26 patients excluded due to GCP violations. Safety set included all randomized patients minus 1 patient who did not receive study drug: 4821 patients
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Valsartan | Total
Number analyzed (Participants) | 2419 | 2403 | 4822
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 415 | 415 | 830
  >=65 years | 2004 | 1988 | 3992
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1247 | 1244 | 2491
  Male | 1172 | 1159 | 2331
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1975 | 1958 | 3933
  Black | 52 | 50 | 102
  Asian | 297 | 310 | 607
  Native American | 28 | 23 | 51
  Pacific Islander | 0 | 1 | 1
  Other | 67 | 61 | 128

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Primary Composite Events of Cardiovascular (CV) Death and Total (First and Recurrent) HF Hospitalizations.
Description: The primary objective of this study is to compare LCZ696 to valsartan in reducing the rate of the composite endpoint of CV death and total (first and recurrent) HF hospitalizations, in HF patients (New York Heart Association [NYHA] Class II-IV) with preserved ejection fraction (left ventricular ejection fraction [LVEF] ≥45%). The treatment arm with the lower rate of events will be deemed as having a successful response.
Time Frame: Total follow up time (up to 57 months)
Population: Full Analysis Set - This was the primary efficacy population applied in efficacy analyses for all efficacy endpoints.
Measure: Number; unit: Events
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 2407 | 2389
Events
  Primary Composite Events | 894 | 1009
  Total Hospitalizations for heart failure | 690 | 797
  Cardiovascular death | 204 | 212
Statistical Analysis 1: Comparison: LCZ696 vs Valsartan; Primary Composite Events; Test type: Superiority; p = 0.0587, Proportional Rates Model (LWYY) — 1-sided p-value 0.0294; Treatment as fixed-effect factor and stratified by region and with robust variance estimate; Rate Ratio = 0.8698, 95% CI 2-sided [0.7526 to 1.0052]
Statistical Analysis 2: Comparison: LCZ696 vs Valsartan; Total Hospitalizations for heart failure; Test type: Superiority; p = 0.0556, Joint Frality Model — 1-sided p-value 0.0278; Treatment and region as fixed-effect factors; Rate Ratio = 0.8511, 95% CI 2-sided [0.7216 to 1.0039]
Statistical Analysis 3: Comparison: LCZ696 vs Valsartan; Cardiovascular Death; Test type: Superiority; p = 0.6241, Cox's proportional hazard model — 1-sided p-value 0.3120; Hazard Ratio (HR) = 0.9531, 95% CI 2-sided [0.7863 to 1.1551]

2. Secondary Outcome: Change in the Clinical Summary Score From Baseline to Month 8 by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The KCCQ is a validated instrument for self-assessment of quality of life and health status in heart failure (HF) patients. The clinical summary score, which is derived from the physical limitations and heart failure (HF) symptoms domains of the KCCQ is a valid measure for assessing the patient's health aspects that may be influenced by CV medications. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. Evaluation of change from baseline to month 8 in KCCQ a most sensitive, specific, and responsive health-related quality of life measure for heart failure symptoms and physical limitations.
Time Frame: Baseline, 8 months
Population: Full Analysis Set-This was the primary efficacy population applied in efficacy analyses for all efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 2407 | 2389
Points on a scale | -1.5073 (0.3709) | -2.5338 (0.3729)
Statistical Analysis 1: Comparison: LCZ696 vs Valsartan; Clinical Summary Score; Test type: Superiority; p = 0.0510, Mixed Models Analysis; Least Squares Mean of Difference = 1.0264, 95% CI 2-sided [-0.0047 to 2.0576]

3. Secondary Outcome: Change From Baseline to Month 8 in New York Heart Association (NYHA) Functional Class
Description: Evaluation of change from baseline to Month 8 in NYHA functional class, a well established grading scale used to classify a heart failure's (HF) patients' level of functionality based on the signs and symptoms of HF exhibited by the patient.
Time Frame: Baseline, 8 months
Population: Full Analysis Set - This was the primary efficacy population applied in efficacy analyses for all efficacy endpoints. However, this endpoint only includes those participants who had assessments completed for both Baseline and Month 8 visits; as that is the only way a change could be calculated and analyzed.
Measure: Number; unit: Number of Participants
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 2407 | 2389
Number of Participants
  Improved (n=2316, 2302): number analyzed (Participants) | 2316 | 2302
  Improved (n=2316, 2302) | 347 | 289
  Unchanged (n=2316, 2302): number analyzed (Participants) | 2316 | 2302
  Unchanged (n=2316, 2302) | 1767 | 1792
  Worsened (n=2316, 2302): number analyzed (Participants) | 2316 | 2302
  Worsened (n=2316, 2302) | 202 | 221
Statistical Analysis 1: Comparison: LCZ696 vs Valsartan; NYHA Class Change; Test type: Superiority; p = 0.0035, Repeated measures cumulative odds model; The response variable is the change from baseline to any scheduled time points up to Month 8; Odds Ratio (OR) = 1.4475, 95% CI 2-sided [1.1294 to 1.8552]

4. Secondary Outcome: Participants With First Occurrence of a Composite Renal Endpoint
Description: Analyis of composite renal endpoint defined as renal death, or reaching ESRD, or ≥50% decline in eGFR relative to baseline, using Cox's proportional hazards model.
Time Frame: Randomization to total follow-up time (up to 57 months)
Population: Full Analysis Set -This was the primary efficacy population applied in efficacy analyses for all efficacy endpoints.
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 2407 | 2389
Participants
  Composite renal endpoint | 33 | 64
  Renal Death | 1 | 1
  Reaching ESRD | 7 | 12
  >=50% decline in eGFR from baseline | 27 | 60
Statistical Analysis 1: Comparison: LCZ696 vs Valsartan; Composite renal endpoint; Test type: Superiority; p = 0.0014, Cox's proportional hazards model; Treatment as fixed factor and stratified by region; Hazard Ratio (HR) = 0.5041, 95% CI 2-sided [0.3312 to 0.7673]
Statistical Analysis 2: Comparison: LCZ696 vs Valsartan; Renal Death; Test type: Superiority; p = 0.9588, Cox's proportional hazards model; Treatment as fixed factor and stratified by region; Hazard Ratio (HR) = 0.9295, 95% CI 2-sided [0.0581 to 14.861]
Statistical Analysis 3: Comparison: LCZ696 vs Valsartan; Reaching ESRD; Test type: Superiority; p = 0.2484, Cox's proportional hazards model; Treatment as fixed factor and stratified by region; Hazard Ratio (HR) = 0.5774, 95% CI 2-sided [0.2272 to 1.4672]
Statistical Analysis 4: Comparison: LCZ696 vs Valsartan; >=50% decline in eGFR from baseline; Test type: Superiority; p = 0.0004, Cox's proportional hazards model; Treatment as fixed factor and stratified by region; Hazard Ratio (HR) = 0.4407, 95% CI 2-sided [0.2798 to 0.6942]

5. Secondary Outcome: All-cause Mortality
Description: Analysis for all-cause mortality using Cox's proportional hazards model.
Time Frame: Randomization to total follow up time (up to 57 months)
Population: Full Analysis Set -This was the primary efficacy population applied in efficacy analyses for all efficacy endpoints.
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 2407 | 2389
Participants | 342 | 349
Statistical Analysis 1: Comparison: LCZ696 vs Valsartan; All-cause mortality; Test type: Superiority; p = 0.6846, Cox's proportional hazards model; Treatment as fixed factor and stratified by region; Hazard Ratio (HR) = 0.9696, 95% CI 2-sided [0.8352 to 1.1255]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approx. 5 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. Safety set included all randomized patients minus 1 patient who did not receive study drug: 4821 patients.
Groups:
- All Patients: Total patients
Arm/Group | LCZ696 | Valsartan | All Patients
All-Cause Mortality (participants affected / at risk) | 347/2419 | 357/2402 | 704/4821
Serious Adverse Events (participants affected / at risk) | 1424/2419 | 1416/2402 | 2840/4821
Other Adverse Events (participants affected / at risk) | 2005/2419 | 1995/2402 | 4000/4821
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=2419) | Valsartan (N=2402) | All Patients (N=4821)
Acquired haemophilia (Blood and lymphatic system disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 68 | 67 | 135
Anaemia macrocytic (Blood and lymphatic system disorders) | 2 | 1 | 3
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 2 | 0 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 7 | 9
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 6 | 11
Leukocytosis (Blood and lymphatic system disorders) | 1 | 6 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 2
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 3 | 1 | 4
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 1
Splenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1 | 7
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 11 | 13 | 24
Acute left ventricular failure (Cardiac disorders) | 14 | 15 | 29
Acute myocardial infarction (Cardiac disorders) | 60 | 54 | 114
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 42 | 50 | 92
Angina unstable (Cardiac disorders) | 50 | 43 | 93
Aortic valve disease (Cardiac disorders) | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 2 | 2 | 4
Aortic valve stenosis (Cardiac disorders) | 4 | 3 | 7
Arrhythmia (Cardiac disorders) | 4 | 4 | 8
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 4 | 8
Atrial fibrillation (Cardiac disorders) | 162 | 145 | 307
Atrial flutter (Cardiac disorders) | 31 | 23 | 54
Atrial tachycardia (Cardiac disorders) | 7 | 2 | 9
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block (Cardiac disorders) | 6 | 4 | 10
Atrioventricular block complete (Cardiac disorders) | 8 | 11 | 19
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 4 | 3 | 7
Bradyarrhythmia (Cardiac disorders) | 3 | 3 | 6
Bradycardia (Cardiac disorders) | 27 | 24 | 51
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 17 | 30 | 47
Cardiac asthma (Cardiac disorders) | 1 | 0 | 1
Cardiac discomfort (Cardiac disorders) | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 340 | 380 | 720
Cardiac failure acute (Cardiac disorders) | 85 | 77 | 162
Cardiac failure chronic (Cardiac disorders) | 26 | 30 | 56
Cardiac failure congestive (Cardiac disorders) | 86 | 83 | 169
Cardiac fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1 | 1
Cardiac tamponade (Cardiac disorders) | 2 | 2 | 4
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 1
Cardiac ventricular disorder (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 15 | 13 | 28
Cardiogenic shock (Cardiac disorders) | 12 | 6 | 18
Cardiomegaly (Cardiac disorders) | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 3 | 3
Cardiopulmonary failure (Cardiac disorders) | 4 | 1 | 5
Cardiorenal syndrome (Cardiac disorders) | 2 | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 3 | 4
Chronic left ventricular failure (Cardiac disorders) | 3 | 1 | 4
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1 | 3
Cor pulmonale (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 24 | 27 | 51
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 5 | 2 | 7
Hypertensive heart disease (Cardiac disorders) | 1 | 3 | 4
Intracardiac mass (Cardiac disorders) | 1 | 1 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 4 | 1 | 5
Left ventricular dysfunction (Cardiac disorders) | 0 | 3 | 3
Left ventricular failure (Cardiac disorders) | 6 | 5 | 11
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Mitral valve calcification (Cardiac disorders) | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 7 | 8 | 15
Mitral valve prolapse (Cardiac disorders) | 2 | 0 | 2
Myocardial infarction (Cardiac disorders) | 32 | 35 | 67
Myocardial ischaemia (Cardiac disorders) | 7 | 11 | 18
Myocardial rupture (Cardiac disorders) | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 2 | 0 | 2
Nodal rhythm (Cardiac disorders) | 0 | 2 | 2
Palpitations (Cardiac disorders) | 3 | 4 | 7
Pericardial effusion (Cardiac disorders) | 3 | 4 | 7
Pericarditis (Cardiac disorders) | 1 | 2 | 3
Pericarditis constrictive (Cardiac disorders) | 1 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 3 | 1 | 4
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 3 | 3
Sinoatrial block (Cardiac disorders) | 0 | 1 | 1
Sinus arrest (Cardiac disorders) | 1 | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 8 | 9
Sinus node dysfunction (Cardiac disorders) | 18 | 12 | 30
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 2
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 6 | 3 | 9
Systolic dysfunction (Cardiac disorders) | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 3 | 0 | 3
Tachycardia (Cardiac disorders) | 3 | 1 | 4
Torsade de pointes (Cardiac disorders) | 1 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 3 | 3
Trifascicular block (Cardiac disorders) | 1 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1
Ventricular dyssynchrony (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 1 | 3
Ventricular fibrillation (Cardiac disorders) | 4 | 5 | 9
Ventricular tachycardia (Cardiac disorders) | 9 | 4 | 13
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 1
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 | 1 | 1
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 1 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 0 | 2
LUMBAR syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 1
Vertebral artery hypoplasia (Congenital, familial and genetic disorders) | 1 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 3 | 9
Vertigo positional (Ear and labyrinth disorders) | 5 | 1 | 6
Vestibular ischaemia (Ear and labyrinth disorders) | 1 | 0 | 1
Goitre (Endocrine disorders) | 0 | 3 | 3
Hypercorticoidism (Endocrine disorders) | 1 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 3 | 6
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 1 | 2
Parathyroid hyperplasia (Endocrine disorders) | 1 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1 | 1
Blindness unilateral (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 14 | 12 | 26
Cataract diabetic (Eye disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 3 | 4
Entropion (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Glaucoma (Eye disorders) | 2 | 1 | 3
Macular degeneration (Eye disorders) | 1 | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 1 | 2
Maculopathy (Eye disorders) | 0 | 1 | 1
Narrow anterior chamber angle (Eye disorders) | 1 | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 1
Pterygium (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 1 | 3 | 4
Retinal haemorrhage (Eye disorders) | 1 | 2 | 3
Retinal vein occlusion (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 3 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 8 | 14
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 7
Abdominal wall haematoma (Gastrointestinal disorders) | 2 | 2 | 4
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 3 | 4
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 8 | 9 | 17
Chronic gastritis (Gastrointestinal disorders) | 2 | 3 | 5
Colitis (Gastrointestinal disorders) | 5 | 3 | 8
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2 | 3
Colitis microscopic (Gastrointestinal disorders) | 2 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 6 | 8
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 | 1 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 14 | 27
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 3 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 2 | 3
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 2
Duodenal polyp (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 3 | 4 | 7
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 3 | 4
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 5
Enteritis (Gastrointestinal disorders) | 3 | 1 | 4
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 2
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 3 | 4
Gastric polyps (Gastrointestinal disorders) | 1 | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 8 | 3 | 11
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 4 | 6
Gastritis (Gastrointestinal disorders) | 3 | 7 | 10
Gastritis erosive (Gastrointestinal disorders) | 1 | 7 | 8
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 29 | 32 | 61
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 7
Haematemesis (Gastrointestinal disorders) | 2 | 1 | 3
Haematochezia (Gastrointestinal disorders) | 4 | 3 | 7
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 5 | 3 | 8
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 3 | 5
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 10 | 13 | 23
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 4
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 3 | 3 | 6
Intestinal obstruction (Gastrointestinal disorders) | 5 | 5 | 10
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 2 | 3
Large intestine polyp (Gastrointestinal disorders) | 5 | 4 | 9
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 6 | 7
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 1 | 2
Melaena (Gastrointestinal disorders) | 7 | 6 | 13
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 5 | 17
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 1 | 3
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 3 | 5
Pancreatitis acute (Gastrointestinal disorders) | 5 | 9 | 14
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 4 | 13
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 1 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 1 | 3
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 5 | 12
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 2 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 11 | 18
Varices oesophageal (Gastrointestinal disorders) | 3 | 2 | 5
Vomiting (Gastrointestinal disorders) | 9 | 11 | 20
Adverse drug reaction (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 12 | 21 | 33
Cardiac death (General disorders) | 3 | 6 | 9
Catheter site haemorrhage (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 4 | 1 | 5
Chest pain (General disorders) | 2 | 1 | 3
Concomitant disease progression (General disorders) | 1 | 0 | 1
Condition aggravated (General disorders) | 1 | 0 | 1
Death (General disorders) | 34 | 23 | 57
Disuse syndrome (General disorders) | 1 | 0 | 1
Euthanasia (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 4 | 4 | 8
Gait disturbance (General disorders) | 3 | 3 | 6
General physical health deterioration (General disorders) | 9 | 5 | 14
Hyperthermia (General disorders) | 0 | 1 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 1
Impaired healing (General disorders) | 3 | 0 | 3
Impaired self-care (General disorders) | 1 | 0 | 1
Implant site haemorrhage (General disorders) | 1 | 0 | 1
Incarcerated hernia (General disorders) | 2 | 0 | 2
Influenza like illness (General disorders) | 1 | 0 | 1
Lithiasis (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 2 | 2 | 4
Mass (General disorders) | 1 | 3 | 4
Medical device discomfort (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 10 | 7 | 17
Necrosis (General disorders) | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 42 | 37 | 79
Oedema (General disorders) | 2 | 0 | 2
Oedema peripheral (General disorders) | 6 | 12 | 18
Pain (General disorders) | 1 | 3 | 4
Peripheral swelling (General disorders) | 1 | 3 | 4
Pyrexia (General disorders) | 8 | 13 | 21
Stenosis (General disorders) | 1 | 0 | 1
Sudden cardiac death (General disorders) | 15 | 16 | 31
Sudden death (General disorders) | 21 | 22 | 43
Surgical failure (General disorders) | 1 | 1 | 2
Swelling (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 5 | 6
Treatment noncompliance (General disorders) | 0 | 1 | 1
Ulcer haemorrhage (General disorders) | 1 | 0 | 1
Unevaluable event (General disorders) | 0 | 3 | 3
Vascular stent stenosis (General disorders) | 1 | 2 | 3
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 5 | 4 | 9
Biliary colic (Hepatobiliary disorders) | 2 | 1 | 3
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 4 | 8
Cholangitis acute (Hepatobiliary disorders) | 1 | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 14 | 11 | 25
Cholecystitis acute (Hepatobiliary disorders) | 8 | 9 | 17
Cholecystitis chronic (Hepatobiliary disorders) | 5 | 2 | 7
Cholelithiasis (Hepatobiliary disorders) | 17 | 19 | 36
Cholelithiasis migration (Hepatobiliary disorders) | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 2
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1 | 1
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder rupture (Hepatobiliary disorders) | 2 | 0 | 2
Haemobilia (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 6 | 10
Hepatic cyst (Hepatobiliary disorders) | 5 | 6 | 11
Hepatic failure (Hepatobiliary disorders) | 3 | 4 | 7
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 5 | 10
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 10 | 10 | 20
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 2 | 2
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 2 | 3
Hepatomegaly (Hepatobiliary disorders) | 0 | 2 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 2 | 3
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 8 | 5 | 13
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 4 | 5
Liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 | 2 | 3
Portal hypertension (Hepatobiliary disorders) | 1 | 2 | 3
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Steatohepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 1
Sarcoidosis (Immune system disorders) | 1 | 1 | 2
Abdominal sepsis (Infections and infestations) | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 1 | 1
Abscess limb (Infections and infestations) | 2 | 0 | 2
Abscess neck (Infections and infestations) | 0 | 1 | 1
Abscess oral (Infections and infestations) | 1 | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 1
Acute endocarditis (Infections and infestations) | 1 | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 3 | 3
Appendicitis (Infections and infestations) | 2 | 4 | 6
Arthritis bacterial (Infections and infestations) | 3 | 6 | 9
Arthritis infective (Infections and infestations) | 0 | 1 | 1
Aspergillus infection (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 6 | 7 | 13
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 1
Bacterial rhinitis (Infections and infestations) | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 2 | 2
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 2 | 2
Biliary sepsis (Infections and infestations) | 0 | 1 | 1
Biliary tract infection (Infections and infestations) | 0 | 1 | 1
Bone abscess (Infections and infestations) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 32 | 41 | 73
Bronchitis viral (Infections and infestations) | 0 | 2 | 2
Campylobacter infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 30 | 25 | 55
Chest wall abscess (Infections and infestations) | 1 | 0 | 1
Cholangitis infective (Infections and infestations) | 2 | 0 | 2
Chronic sinusitis (Infections and infestations) | 1 | 0 | 1
Clostridium colitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 6 | 3 | 9
Clostridium difficile infection (Infections and infestations) | 3 | 2 | 5
Colonic abscess (Infections and infestations) | 1 | 2 | 3
Complicated appendicitis (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 2 | 1 | 3
Cystitis bacterial (Infections and infestations) | 1 | 0 | 1
Cystitis escherichia (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 2
Dengue fever (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 2 | 1 | 3
Diabetic foot infection (Infections and infestations) | 1 | 2 | 3
Diabetic gangrene (Infections and infestations) | 0 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 9 | 12
Eczema infected (Infections and infestations) | 1 | 1 | 2
Embolic pneumonia (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 2 | 3 | 5
Enteritis infectious (Infections and infestations) | 1 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 11 | 7 | 18
Escherichia bacteraemia (Infections and infestations) | 0 | 2 | 2
Escherichia sepsis (Infections and infestations) | 1 | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 3
Gangrene (Infections and infestations) | 3 | 3 | 6
Gastroenteritis (Infections and infestations) | 21 | 16 | 37
Gastroenteritis bacterial (Infections and infestations) | 0 | 2 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 1 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 2 | 2
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 3
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1
Genital herpes zoster (Infections and infestations) | 0 | 1 | 1
Haematoma infection (Infections and infestations) | 1 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 4 | 6
Hordeolum (Infections and infestations) | 0 | 1 | 1
Human anaplasmosis (Infections and infestations) | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 2 | 4 | 6
Infection (Infections and infestations) | 1 | 3 | 4
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 2 | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 3 | 5
Influenza (Infections and infestations) | 16 | 11 | 27
Intervertebral discitis (Infections and infestations) | 1 | 2 | 3
Intestinal sepsis (Infections and infestations) | 0 | 1 | 1
Intracranial infection (Infections and infestations) | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 2 | 0 | 2
Labyrinthitis (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1
Liver abscess (Infections and infestations) | 0 | 2 | 2
Localised infection (Infections and infestations) | 4 | 5 | 9
Lower respiratory tract infection (Infections and infestations) | 11 | 12 | 23
Lower respiratory tract infection viral (Infections and infestations) | 1 | 1 | 2
Lung abscess (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 12 | 11 | 23
Lymphangitis (Infections and infestations) | 0 | 1 | 1
Mediastinitis (Infections and infestations) | 0 | 2 | 2
Medical device site infection (Infections and infestations) | 1 | 0 | 1
Meningitis enterococcal (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 2
Orchitis (Infections and infestations) | 1 | 1 | 2
Osteomyelitis (Infections and infestations) | 7 | 3 | 10
Otitis media (Infections and infestations) | 0 | 1 | 1
Pelvic abscess (Infections and infestations) | 1 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 2 | 2
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 3 | 0 | 3
Pneumonia (Infections and infestations) | 162 | 178 | 340
Pneumonia bacterial (Infections and infestations) | 4 | 5 | 9
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia viral (Infections and infestations) | 2 | 1 | 3
Post procedural infection (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 3 | 3 | 6
Pseudomembranous colitis (Infections and infestations) | 1 | 2 | 3
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 3 | 3 | 6
Pyelonephritis acute (Infections and infestations) | 4 | 3 | 7
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 2 | 3
Respiratory tract infection (Infections and infestations) | 19 | 21 | 40
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 3
Salmonellosis (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 34 | 37 | 71
Septic encephalopathy (Infections and infestations) | 0 | 1 | 1
Septic necrosis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 21 | 16 | 37
Severe acute respiratory syndrome (Infections and infestations) | 0 | 1 | 1
Shunt infection (Infections and infestations) | 0 | 1 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 3 | 3
Staphylococcal infection (Infections and infestations) | 1 | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 2
Streptococcal bacteraemia (Infections and infestations) | 1 | 1 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 3 | 3
Syphilis (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Tracheobronchitis (Infections and infestations) | 2 | 2 | 4
Tuberculosis (Infections and infestations) | 0 | 1 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 11
Urethritis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 54 | 68 | 122
Urosepsis (Infections and infestations) | 11 | 14 | 25
Vestibular neuronitis (Infections and infestations) | 2 | 1 | 3
Viral infection (Infections and infestations) | 1 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Wound abscess (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 2 | 3 | 5
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 3 | 3
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1 | 2
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2 | 2
Anastomotic ulcer (Injury, poisoning and procedural complications) | 2 | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 7 | 4 | 11
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 3 | 7
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 4 | 7
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Extra dose administered (Injury, poisoning and procedural complications) | 1 | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 33 | 26 | 59
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 8 | 13
Femur fracture (Injury, poisoning and procedural complications) | 11 | 20 | 31
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 5 | 6 | 11
Hip fracture (Injury, poisoning and procedural complications) | 13 | 14 | 27
Humerus fracture (Injury, poisoning and procedural complications) | 5 | 7 | 12
Hypobarism (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2 | 3
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 3 | 5
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 4 | 1 | 5
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 2 | 5
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 4 | 2 | 6
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 3
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 7 | 1 | 8
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 11 | 6 | 17
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sedation complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 6 | 2 | 8
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 8 | 11
Spinal fracture (Injury, poisoning and procedural complications) | 6 | 2 | 8
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Stomal hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 7 | 8 | 15
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2 | 4
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 8 | 10
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 2
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 2 | 4
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 3 | 4
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 4
Anticoagulation drug level above therapeutic (Investigations) | 2 | 4 | 6
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 6
Bleeding time abnormal (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 4 | 5
Blood glucose abnormal (Investigations) | 1 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 1
Blood glucose fluctuation (Investigations) | 2 | 0 | 2
Blood glucose increased (Investigations) | 1 | 2 | 3
Blood osmolarity decreased (Investigations) | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 2 | 1 | 3
Blood sodium decreased (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 1 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 1
Cardiac output decreased (Investigations) | 1 | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1 | 1
General physical condition abnormal (Investigations) | 0 | 1 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 3 | 3
Haemoglobin decreased (Investigations) | 0 | 3 | 3
Heart rate decreased (Investigations) | 0 | 1 | 1
Heart rate irregular (Investigations) | 1 | 1 | 2
Hepatic enzyme increased (Investigations) | 7 | 6 | 13
Inflammatory marker increased (Investigations) | 0 | 2 | 2
Influenza virus test positive (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 3 | 2 | 5
Lipase increased (Investigations) | 0 | 1 | 1
Myocardial necrosis marker increased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Precancerous cells present (Investigations) | 1 | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0 | 1
Pulse absent (Investigations) | 1 | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 2 | 3
Troponin I increased (Investigations) | 0 | 1 | 1
Troponin T increased (Investigations) | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 4 | 4
Urine output decreased (Investigations) | 0 | 1 | 1
Ventilation/perfusion scan abnormal (Investigations) | 1 | 0 | 1
Visual field tests abnormal (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 2
Cachexia (Metabolism and nutrition disorders) | 2 | 1 | 3
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 18 | 26 | 44
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 8 | 17
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 3 | 7
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 3 | 9 | 12
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 8 | 8 | 16
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 5 | 11 | 16
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 16 | 26
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 19 | 42 | 61
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 20 | 6 | 26
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 14 | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 17 | 34
Hypoosmolar state (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 4 | 1 | 5
Iron deficiency (Metabolism and nutrition disorders) | 0 | 4 | 4
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 3 | 3
Marasmus (Metabolism and nutrition disorders) | 1 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 3 | 6
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 8 | 13
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 22
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
CREST syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 | 5 | 14
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myositis ossificans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 31 | 28 | 59
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 8
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 | 3 | 9
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 10
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 9
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 6 | 11
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 7
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 11 | 22
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 7
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Breast angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8 | 14
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 5
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 9
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 7
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 7
Hormone-refractory prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 5
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 4
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10 | 18
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6 | 13
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 7
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 6
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 | 15
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 5
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4 | 10
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8 | 14
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 5
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 4
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Vaginal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 1 | 4 | 5
Ataxia (Nervous system disorders) | 0 | 1 | 1
Brain hypoxia (Nervous system disorders) | 1 | 1 | 2
Brain injury (Nervous system disorders) | 1 | 1 | 2
Brain oedema (Nervous system disorders) | 2 | 1 | 3
Brain stem stroke (Nervous system disorders) | 0 | 1 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 2 | 2
Carotid artery disease (Nervous system disorders) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 9 | 7 | 16
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 1
Cerebellar haematoma (Nervous system disorders) | 0 | 1 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 2 | 2
Cerebellar ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 5 | 6 | 11
Cerebral infarction (Nervous system disorders) | 17 | 18 | 35
Cerebral ischaemia (Nervous system disorders) | 3 | 3 | 6
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 39 | 42 | 81
Cerebrovascular disorder (Nervous system disorders) | 1 | 1 | 2
Cerebrovascular insufficiency (Nervous system disorders) | 2 | 1 | 3
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 7 | 2 | 9
Coma (Nervous system disorders) | 1 | 4 | 5
Dementia (Nervous system disorders) | 2 | 1 | 3
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1 | 2
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 17 | 11 | 28
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 5 | 4 | 9
Encephalopathy (Nervous system disorders) | 1 | 6 | 7
Epilepsy (Nervous system disorders) | 0 | 3 | 3
Facial paralysis (Nervous system disorders) | 2 | 0 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 1 | 2
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 2 | 1 | 3
Haemorrhagic stroke (Nervous system disorders) | 3 | 3 | 6
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 3 | 10 | 13
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 1 | 2
Hepatic encephalopathy (Nervous system disorders) | 1 | 5 | 6
Hydrocephalus (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 3
Hypoglycaemic coma (Nervous system disorders) | 1 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 2 | 1 | 3
Intracranial haematoma (Nervous system disorders) | 0 | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 32 | 29 | 61
Lacunar infarction (Nervous system disorders) | 4 | 2 | 6
Lacunar stroke (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 1 | 3
Loss of consciousness (Nervous system disorders) | 3 | 3 | 6
Lumbar radiculopathy (Nervous system disorders) | 1 | 2 | 3
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 6 | 3 | 9
Migraine (Nervous system disorders) | 1 | 0 | 1
Mixed dementia (Nervous system disorders) | 0 | 1 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 1
Movement disorder (Nervous system disorders) | 1 | 0 | 1
Multiple system atrophy (Nervous system disorders) | 1 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 1
Myasthenic syndrome (Nervous system disorders) | 1 | 0 | 1
Myelopathy (Nervous system disorders) | 2 | 0 | 2
Myoclonus (Nervous system disorders) | 1 | 1 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 2 | 1 | 3
Parkinsonism (Nervous system disorders) | 0 | 2 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 1
Post stroke epilepsy (Nervous system disorders) | 1 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 3 | 3 | 6
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 2 | 2 | 4
Resting tremor (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 4 | 4 | 8
Seizure (Nervous system disorders) | 6 | 2 | 8
Sensory disturbance (Nervous system disorders) | 2 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 2 | 2
Speech disorder (Nervous system disorders) | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1
Spinal cord disorder (Nervous system disorders) | 0 | 1 | 1
Spondylitic myelopathy (Nervous system disorders) | 2 | 0 | 2
Status epilepticus (Nervous system disorders) | 0 | 2 | 2
Stroke in evolution (Nervous system disorders) | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 4 | 7
Syncope (Nervous system disorders) | 41 | 57 | 98
Thalamus haemorrhage (Nervous system disorders) | 0 | 1 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 34 | 26 | 60
Tremor (Nervous system disorders) | 0 | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 1 | 0 | 1
VIth nerve paresis (Nervous system disorders) | 1 | 0 | 1
Vascular dementia (Nervous system disorders) | 2 | 2 | 4
Vascular parkinsonism (Nervous system disorders) | 0 | 1 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 2 | 6
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 1
Device battery issue (Product Issues) | 1 | 2 | 3
Device breakage (Product Issues) | 1 | 0 | 1
Device damage (Product Issues) | 1 | 0 | 1
Device defective (Product Issues) | 0 | 2 | 2
Device dislocation (Product Issues) | 2 | 2 | 4
Device failure (Product Issues) | 0 | 1 | 1
Device leakage (Product Issues) | 0 | 1 | 1
Device loosening (Product Issues) | 0 | 1 | 1
Device malfunction (Product Issues) | 1 | 1 | 2
Device occlusion (Product Issues) | 0 | 1 | 1
Lead dislodgement (Product Issues) | 1 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 1
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 3
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 1
Behaviour disorder (Psychiatric disorders) | 0 | 1 | 1
Completed suicide (Psychiatric disorders) | 4 | 2 | 6
Confusional state (Psychiatric disorders) | 6 | 7 | 13
Delirium (Psychiatric disorders) | 7 | 11 | 18
Delirium febrile (Psychiatric disorders) | 0 | 1 | 1
Delusion (Psychiatric disorders) | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 6 | 7 | 13
Disorientation (Psychiatric disorders) | 1 | 1 | 2
Hallucination (Psychiatric disorders) | 2 | 1 | 3
Major depression (Psychiatric disorders) | 1 | 2 | 3
Mental disorder (Psychiatric disorders) | 1 | 1 | 2
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 5 | 8
Organic brain syndrome (Psychiatric disorders) | 1 | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0 | 1
Personality disorder (Psychiatric disorders) | 1 | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 90 | 110 | 200
Anuria (Renal and urinary disorders) | 2 | 0 | 2
Azotaemia (Renal and urinary disorders) | 3 | 3 | 6
Bladder diverticulum (Renal and urinary disorders) | 0 | 1 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 13 | 14 | 27
Dysuria (Renal and urinary disorders) | 0 | 2 | 2
End stage renal disease (Renal and urinary disorders) | 3 | 3 | 6
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 1
Glomerulonephropathy (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 8 | 13
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 3 | 5
Nephrolithiasis (Renal and urinary disorders) | 3 | 5 | 8
Nephropathy toxic (Renal and urinary disorders) | 0 | 3 | 3
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1 | 2
Oliguria (Renal and urinary disorders) | 0 | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 3 | 4
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 2 | 2
Renal disorder (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 31 | 29 | 60
Renal impairment (Renal and urinary disorders) | 24 | 48 | 72
Renal infarct (Renal and urinary disorders) | 3 | 0 | 3
Renal injury (Renal and urinary disorders) | 0 | 2 | 2
Renal mass (Renal and urinary disorders) | 0 | 1 | 1
Renal pain (Renal and urinary disorders) | 1 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 3 | 3
Renal vein stenosis (Renal and urinary disorders) | 1 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 4
Urinary retention (Renal and urinary disorders) | 8 | 8 | 16
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | 2
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 5 | 13
Breast calcifications (Reproductive system and breast disorders) | 0 | 1 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Endometrial thickening (Reproductive system and breast disorders) | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1 | 3
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 2
Scrotal inflammation (Reproductive system and breast disorders) | 1 | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 1 | 2
Uterine prolapse (Reproductive system and breast disorders) | 2 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 26
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 20 | 24 | 44
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 19
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 42 | 67 | 109
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 64 | 106
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 9
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 8
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 32
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Presbyphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 33
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 13
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 23
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29 | 32 | 61
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 9
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 5 | 1 | 6
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 5 | 7
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rhinophyma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 | 3 | 8
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Immobile (Social circumstances) | 1 | 0 | 1
Living in residential institution (Social circumstances) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 2 | 2
Angiopathy (Vascular disorders) | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 2 | 8 | 10
Aortic aneurysm rupture (Vascular disorders) | 2 | 1 | 3
Aortic dissection (Vascular disorders) | 0 | 1 | 1
Aortic rupture (Vascular disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 13 | 12 | 25
Aortic thrombosis (Vascular disorders) | 1 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 2 | 1 | 3
Arteriosclerosis (Vascular disorders) | 1 | 1 | 2
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 2 | 2
Circulatory collapse (Vascular disorders) | 3 | 2 | 5
Deep vein thrombosis (Vascular disorders) | 4 | 7 | 11
Dry gangrene (Vascular disorders) | 1 | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 1 | 2
Extremity necrosis (Vascular disorders) | 2 | 0 | 2
Haematoma (Vascular disorders) | 7 | 8 | 15
Haemorrhage (Vascular disorders) | 2 | 1 | 3
Haemorrhagic infarction (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 16 | 25 | 41
Hypertensive crisis (Vascular disorders) | 4 | 8 | 12
Hypertensive emergency (Vascular disorders) | 1 | 3 | 4
Hypertensive urgency (Vascular disorders) | 6 | 1 | 7
Hypotension (Vascular disorders) | 52 | 47 | 99
Hypovolaemic shock (Vascular disorders) | 1 | 2 | 3
Iliac artery embolism (Vascular disorders) | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 2 | 1 | 3
Ischaemia (Vascular disorders) | 0 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 1
Leriche syndrome (Vascular disorders) | 1 | 1 | 2
Lymphoedema (Vascular disorders) | 0 | 4 | 4
Orthostatic hypertension (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 5 | 9 | 14
Peripheral arterial occlusive disease (Vascular disorders) | 18 | 7 | 25
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 2 | 2 | 4
Peripheral artery stenosis (Vascular disorders) | 3 | 4 | 7
Peripheral artery thrombosis (Vascular disorders) | 2 | 2 | 4
Peripheral coldness (Vascular disorders) | 1 | 0 | 1
Peripheral embolism (Vascular disorders) | 3 | 3 | 6
Peripheral ischaemia (Vascular disorders) | 8 | 7 | 15
Peripheral vascular disorder (Vascular disorders) | 5 | 2 | 7
Peripheral venous disease (Vascular disorders) | 2 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 1
Shock (Vascular disorders) | 0 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 5 | 7
Subclavian artery stenosis (Vascular disorders) | 1 | 1 | 2
Subclavian artery thrombosis (Vascular disorders) | 1 | 0 | 1
Temporal arteritis (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1 | 2
Varicose ulceration (Vascular disorders) | 0 | 2 | 2
Venous thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=2419) | Valsartan (N=2402) | All Patients (N=4821)
Anaemia (Blood and lymphatic system disorders) | 166 | 214 | 380
Angina pectoris (Cardiac disorders) | 87 | 82 | 169
Atrial fibrillation (Cardiac disorders) | 248 | 239 | 487
Bradycardia (Cardiac disorders) | 53 | 85 | 138
Cardiac failure (Cardiac disorders) | 225 | 269 | 494
Palpitations (Cardiac disorders) | 62 | 56 | 118
Vertigo (Ear and labyrinth disorders) | 77 | 60 | 137
Cataract (Eye disorders) | 84 | 70 | 154
Abdominal pain (Gastrointestinal disorders) | 53 | 54 | 107
Constipation (Gastrointestinal disorders) | 100 | 86 | 186
Diarrhoea (Gastrointestinal disorders) | 177 | 180 | 357
Nausea (Gastrointestinal disorders) | 93 | 87 | 180
Vomiting (Gastrointestinal disorders) | 70 | 58 | 128
Asthenia (General disorders) | 60 | 58 | 118
Fatigue (General disorders) | 98 | 107 | 205
Non-cardiac chest pain (General disorders) | 98 | 92 | 190
Oedema peripheral (General disorders) | 166 | 183 | 349
Pyrexia (General disorders) | 59 | 54 | 113
Bronchitis (Infections and infestations) | 177 | 197 | 374
Cellulitis (Infections and infestations) | 61 | 41 | 102
Influenza (Infections and infestations) | 110 | 109 | 219
Nasopharyngitis (Infections and infestations) | 207 | 177 | 384
Pneumonia (Infections and infestations) | 100 | 97 | 197
Respiratory tract infection (Infections and infestations) | 48 | 60 | 108
Upper respiratory tract infection (Infections and infestations) | 145 | 139 | 284
Urinary tract infection (Infections and infestations) | 243 | 268 | 511
Contusion (Injury, poisoning and procedural complications) | 57 | 72 | 129
Fall (Injury, poisoning and procedural complications) | 106 | 90 | 196
Blood creatinine increased (Investigations) | 63 | 65 | 128
Glomerular filtration rate decreased (Investigations) | 85 | 93 | 178
Weight decreased (Investigations) | 71 | 82 | 153
Diabetes mellitus (Metabolism and nutrition disorders) | 52 | 62 | 114
Gout (Metabolism and nutrition disorders) | 76 | 88 | 164
Hyperkalaemia (Metabolism and nutrition disorders) | 238 | 298 | 536
Hyperuricaemia (Metabolism and nutrition disorders) | 62 | 75 | 137
Hypokalaemia (Metabolism and nutrition disorders) | 110 | 100 | 210
Arthralgia (Musculoskeletal and connective tissue disorders) | 152 | 153 | 305
Back pain (Musculoskeletal and connective tissue disorders) | 149 | 170 | 319
Muscle spasms (Musculoskeletal and connective tissue disorders) | 36 | 49 | 85
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 63 | 58 | 121
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 92 | 92 | 184
Pain in extremity (Musculoskeletal and connective tissue disorders) | 81 | 75 | 156
Dizziness (Nervous system disorders) | 229 | 192 | 421
Headache (Nervous system disorders) | 114 | 126 | 240
Syncope (Nervous system disorders) | 42 | 62 | 104
Depression (Psychiatric disorders) | 68 | 70 | 138
Insomnia (Psychiatric disorders) | 75 | 54 | 129
Acute kidney injury (Renal and urinary disorders) | 64 | 65 | 129
Chronic kidney disease (Renal and urinary disorders) | 33 | 50 | 83
Haematuria (Renal and urinary disorders) | 71 | 77 | 148
Renal failure (Renal and urinary disorders) | 85 | 108 | 193
Renal impairment (Renal and urinary disorders) | 287 | 331 | 618
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 57 | 68 | 125
Cough (Respiratory, thoracic and mediastinal disorders) | 188 | 146 | 334
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 217 | 236 | 453
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 42 | 71 | 113
Pruritus (Skin and subcutaneous tissue disorders) | 46 | 51 | 97
Hypertension (Vascular disorders) | 225 | 314 | 539
Hypotension (Vascular disorders) | 529 | 379 | 908

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT01920711/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT01920711/SAP_001.pdf